CLINICAL TRIAL: NCT05204537
Title: The Role of Surgery in Patients With COVID-19 Related Thoracic Complications
Brief Title: The Role of Surgery in Patients With Coronavirus Disease - 19 (COVID-19) Related Thoracic Complications
Acronym: SThor-CoV-2
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Sponsor
Other Study IDs: 3822
Record Dates: First submitted 2022-01-21; First posted 2022-01-24 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Surgical Complication; COVID-19; Pneumothorax; Empyema, Pleural; Abscess; Hemothorax; Thoracic
Keywords: COVID-19, complications, thoracic surgery, mortality
MeSH Terms: conditions — COVID-19; Pneumothorax; Empyema, Pleural; Abscess; Hemothorax | interventions — Cerebral Decortication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who developed in-hospital COVID-19 thoracic complications, surgically managed.: The study population consists of patients who have been surgically treated for COVID-19 thoracic complications.
  Thoracic complications have been defined as any condition involving the thorax, directly or indirectly consequence of COVID-19, including either pathologies strictly related to the infection, or iatrogenic effects of therapeutic attempts to treat it. Since the wide span of diagnosis, the novelty of this pathology and the different protocols adopted by participating centers, it is not possible to identify common criteria for surgical indications. A wide variety of pleuro/parenchimal surgical procedures are included. Patients undergone chest tube placement alone are not included in the study.
  Interventions: Procedure: Lung parenchyma resection; Procedure: Empyemectomy

INTERVENTIONS:
Procedure: Lung parenchyma resection — Lung parenchyma removal
  Other Names: Lobectomy/segmentectomy/pneumonectomy
Procedure: Empyemectomy — Intrapleural cavity effusion removal, parietal pleura removal.
  Other Names: Decortication

SUMMARY:
Thoracic complications directly or indirectly consequence of Coronavirus Disease 2019 (COVID-19) (including either pathologies strictly related to the infection, or iatrogenic effects of therapeutic attempts to treat it) have been described during the pandemic.

Many of the above conditions often require a surgical approach but, based on published data reporting high early postoperative morbidity and mortality, many experts initially advised against any referral to surgery in COVID-19 patients.

Therefore, the issue is if salvage surgical approach should be always excluded or could be considered when it represents the only remaining effective option. In the absence of solid data and recommendations, this is a demanding challenge for thoracic surgeons.

The investigators have coordinated a multicenter study to collect the experience of several worldwide high-volume thoracic surgery departments. Their objective is to investigate efficacy and safety of surgery in COVID-19 patients who developed thoracic complications that required operative management.

DETAILED DESCRIPTION:
The year of 2019 has been characterized by the rise of a new respiratory infection named "severe acute respiratory syndrome coronavirus 2" (Sars-CoV-2). It has rapidly diffused over the world. By November 2021, there were more than 252.000.000 confirmed cases and more than 5.000.000 death worldwide.

A significant amount of effort has been exerted to better understand its optimal management. Mild COVID-19 disease condition can cause symptoms such as fever, cough and shortness of breath as well as tiredness, muscle aches. Yet severe and critical disease state are characterized by dramatic and life-threatening symptoms. Among those, the most common is pneumonia which quickly progress to Acute respiratory distress syndrome (ARDS). Pneumatoceles, parenchymal air-filled cysts, seem to occur more likely in COVID-19 patients as well. The second critical point is blood hypercoagulability, probably due to vascular endothelial cell injury, which is manifested by a higher incidence of venous and arterial thrombosis and pulmonary embolism requiring prolonged anticoagulant prophylactic treatment; these conditions can conspire to unexpected intrapleural bleeding. Moreover, these patients often develop co-infections which lead to further complications such as empyema and septic shock. The above conditions often require a surgical approach but, based on published data reporting high early postoperative morbidity and mortality, many experts initially advised against any referral to surgery in COVID-19 patients.

Therefore, the issue is if salvage surgical approach should be always excluded or could be considered when it represents the only remaining effective option. In the absence of solid data and recommendations, this is a demanding challenge for thoracic surgeons.

Investigators have coordinated a multicenter study to collect the experience of several worldwide high-volume thoracic surgery departments. Their objective is to investigate efficacy and safety of surgery in COVID-19 patients who developed thoracic complications that required operative management. Their first aim is to estimate postoperative survival at 30 days, other endpoints are: postoperative complications incidence and prognostic factors for 30 days mortality and morbidity.

The investigators have designed an observational retrospective multicenter international study, involving nine experienced thoracic surgery departments, in five different countries.

This study has been approved by the research ethics committee at the lead centre and has been conducted in accordance with the Declaration of Helsinki. At the other centers, local principal investigators have been asked with getting approvals.

The study population consists of patients who developed in-hospital COVID-19 thoracic complications, surgically managed from March 2020 to May 2021.

Thoracic complication are defined as any condition involving the thorax, directly or indirectly consequence of COVID-19, including either pathologies strictly related to the infection, or iatrogenic effects of therapeutic attempts to treat it. A wide variety of surgical procedures have been included. Patients undergone chest tube placement alone are not included in the study.

Data are retrospectively collected and entered into a dedicated password-protected database. Demographic, anamnestic, clinical, surgical and outcome-related variables are derived from medical and nursing records, laboratory reports, radiological findings. Patients will be followed up to discharge or to 30 days after surgery if discharge occurred before. Follow up consists of an outpatient clinic visit, including physical examination and chest X-Ray; patients discharged with long-COVID, who are under quarantine at home, according to the regulations in force, are tele medically evaluated.

Primary end-point is postoperative survival at 30 days from surgery. Secondary end-points are postoperative complications. Postoperative complications are graded according to the Thoracic Morbidity and Mortality Classification System from grade I (no need for treatment or intervention) to grade V (leading to death).

The target sample size of about 80 subjects has been derived in order to estimate survival at 30 days post-surgery with a precision of 0.194 (total width of the 95% confidence interval) assuming a survival of 0.77. Baseline characteristics of patients will be described as median (I and III quartiles) and frequencies (percentage). Cumulative incidence of in-hospital mortality and discharge will be estimated by the Aalen-Johansen estimator. Overall mortality at 30 days are obtained by Kaplan-Meier and compared among groups by the log-rank test. In order to account for time to death a multivariable Cox regression model has been applied to identify the variables associated with mortality 30 days after surgery. A multivariable logistic model will be applied to identify variables associated with post-operative complications. The variables included in the models are clinical parameters (age, sex, maximum ventilator support) with the addition of the variables associated with outcomes in the unadjusted analyses (renal insufficiency, pulmonary hypertension, complications surgically treated classified as infective affection (eg. empyema/pneumatoceles) compared to others (eg. pneumothorax, hemothorax, etc.) and type of surgery). Results are presented by hazard ratios (HR) and odds ratios (OR) with 95% confidence intervals (CI). Data will be analyzed using R software (version 4.0.3).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old;
* molecular diagnosis of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection through nose-pharyngeal swab or bronchoalveolar lavage via real-time polymerase chain reaction (PCR) analysis;
* hospital admission because of clinical/radiological diagnosis of pneumonia;
* onset of thoracic complications during hospitalization or prolonged hospitalization requiring thoracic surgical procedures;
* hospital admission from 01/03/2020 to 31/05/2021.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who developed in-hospital COVID-19 thoracic complications, surgically managed in 9 different thoracic surgery department.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Postoperative survival | day 30
  Overall survival at 30 days from surgery

SECONDARY OUTCOMES:
Postoperative complications | 30 days from surgery
  Postoperative complications were graded according to the Thoracic Morbidity and Mortality Classification System from grade I (no need for treatment or intervention) to grade V (leading to death)

CONTACTS AND LOCATIONS:
Overall Officials: Federico Raveglia, MD, Principal Investigator — ASST-Monza
Locations (9):
- Thoracic Surgery, NYU Langone Health, New York, New York, United States
- Thoracic Surgery, Hospital Federal do Andaraí, Rio de Janeiro, Brazil
- India (2):
  - Sunrise hospital., Kochi
  - Thoracic Surgery, Sir Ganga Ram Hospital, New Delhi
- Italy (4):
  - Thoracic Surgery, ASST Spedali Civili, Brescia
  - San Gerardo Hospital, Monza
  - Thoracic Surgery, San Camillo Forlanini Hospital., Roma
  - Thoracic Surgery, San Giovanni Battista Molinette Hospital, Turin
- Thoracic Surgery, University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McGuinness G, Zhan C, Rosenberg N, Azour L, Wickstrom M, Mason DM, Thomas KM, Moore WH. Increased Incidence of Barotrauma in Patients with COVID-19 on Invasive Mechanical Ventilation. Radiology. 2020 Nov;297(2):E252-E262. doi: 10.1148/radiol.2020202352. Epub 2020 Jul 2. PMID 32614258
- [Background] Hamad AM, El-Saka HA. Post COVID-19 large pneumatocele: clinical and pathological perspectives. Interact Cardiovasc Thorac Surg. 2021 Jul 26;33(2):322-324. doi: 10.1093/icvts/ivab072. PMID 33764376
- [Background] Knisely A, Zhou ZN, Wu J, Huang Y, Holcomb K, Melamed A, Advincula AP, Lalwani A, Khoury-Collado F, Tergas AI, St Clair CM, Hou JY, Hershman DL, D'Alton ME, Huang YY, Wright JD. Perioperative Morbidity and Mortality of Patients With COVID-19 Who Undergo Urgent and Emergent Surgical Procedures. Ann Surg. 2021 Jan 1;273(1):34-40. doi: 10.1097/SLA.0000000000004420. PMID 33074900
- [Background] COVIDSurg Collaborative. Mortality and pulmonary complications in patients undergoing surgery with perioperative SARS-CoV-2 infection: an international cohort study. Lancet. 2020 Jul 4;396(10243):27-38. doi: 10.1016/S0140-6736(20)31182-X. Epub 2020 May 29. PMID 32479829
- [Background] Scarci M, Raveglia F, Bortolotti L, Benvenuti M, Merlo L, Petrella L, Cardillo G, Rocco G. COVID-19 After Lung Resection in Northern Italy. Semin Thorac Cardiovasc Surg. 2022 Summer;34(2):726-732. doi: 10.1053/j.semtcvs.2021.03.038. Epub 2021 May 11. PMID 33989754
- [Result] Chang SH, Chen D, Paone D, Geraci TC, Scheinerman J, Bizekis C, Zervos M, Cerfolio RJ. Thoracic surgery outcomes for patients with Coronavirus Disease 2019. J Thorac Cardiovasc Surg. 2021 Dec;162(6):1654-1664. doi: 10.1016/j.jtcvs.2021.01.069. Epub 2021 Jan 30. PMID 33642100

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT05204537/Prot_SAP_000.pdf